CLINICAL TRIAL: NCT01368627
Title: A Prospective, Multinational Investigation of the Supralimus® Sirolimus-Eluting Stent for the Treatment of Unselected Patients With Coronary Lesions in the "Real- World" Clinical Practice
Brief Title: The E-SERIES Registry for Supralimus® Coronary Stent for the Treatment of Unselected Patients With Coronary Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: Cardiovascular Research Center, Brazil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Restenosis; Stent thrombosis; Coronary stents; Angioplasty; Drug Eluting Stents(DES)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supralimus® Sirolimus-Eluting Coronary Stent (Experimental)
  Interventions: Device: Supralimus® Sirolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: Supralimus® Sirolimus-Eluting Coronary Stent — Supralimus® Coronary Stent System consisting of the MATRIX® Coronary Stent having Sirolimus eluting from Biodegradable Polymeric Matrix on a Stainless Steel Platform, Drug concentration 1.4 µg/mm2
  Other Names: Drug Eluting Stent (DES)

SUMMARY:
E-SERIES Registry evaluate the procedural and clinical outcomes of the Supralimus® SES in the treatment of unselected, high risk patients having coronary Artery blockage in the real world clinical practice.

DETAILED DESCRIPTION:
E-SERIES Registry is Prospective, multinational (Asia, South America and Europe), non-randomized, post-marketing web-based registry.

For this Study Up to 100 clinical sites in Asia, South America and Europe. Patients "ALL COMERS" assigned for percutaneous coronary interventions who present with at least one angiographically documented coronary artery lesion suitable for percutaneous treatment with the Supralimus® SES.

All subjects who provided signed informed consent prior to procedure, and have at least one lesion in a major epicardial vessel or major branch (>2.25mm), and are suitable for percutaneous treatment including stenting procedure with the Supralimus® SES. There are no limit regarding the number of lesions and/or study stents to be used, and stenting technique will be left at the operator's discretion; however, it is recommended according to the BEST interventional practice according to the current guidelines.

All patients will undergo follow-up clinical evaluation at 1, 6, 12 and 24 months. Angiographic follow-up will be performed at 6 months in a subset of high risk lesions including bifurcations (first 100 lesions) and left main stem (first 100 lesions).

ELIGIBILITY:
Inclusion Criteria:

1. CLINICAL INCLUSION CRITERIA: Patients >18 years, clinical indication for elective or emergency percutaneous coronary intervention with stent implantation of at least one angiographically documented coronary artery lesion; agreement to undergo ALL study protocol follow-ups.
2. ANGIOGRAPHIC INCLUSION CRITERIA: Diseased coronary vessels with at least one lesion with ≥50% diameter stenosis by visual estimation in a major epicardial vessel or a major branch (>2.25mm) with anatomy suitable for percutaneous treatment with the Supralimus SES.

Exclusion Criteria:

1. CLINICAL EXCLUSION CRITERIA: Known illness with life expectancy <12 months; impossibility to comply with all protocol follow-ups.
2. ANGIOGRAPHIC EXCLUSION CRITERIA: Anatomy unsuitable for percutaneous treatment with implantation of the Supralimus SES.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1274 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
MAJOR ADVERSE CARDIAC EVENTS (MACE) | 12 months

SECONDARY OUTCOMES:
Rates of procedural success | 24 month
Rates of Major Adverse Cardiac Event (MACE) | In-hospital, 30 days, 6 and 24 months
Rates of target lesion revascularization (TLR) | 6 and 12 months
Rates of stent thrombosis (acute, sub-acute, late and very-late) | Up to 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid,, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia São Paulo, SP, Brazil
Locations (7):
- Brazil (7):
  - CIAS- Unimed Vitória, Vitória, Espírito Santo
  - Centro de Cardiologia e Radiologia, Goiânia, Goiás
  - Hospital Luxemburgo, Belo Horizonte, Minas Gerais
  - Hospital Monte Sinai, Juiz de Fora, Minas Gerais
  - Hospital Vita, Curitiba, Paraná
  - H.C.Unesp, Botucatu, São Paulo
  - Hospital São Camilo, São Paulo, São Paulo